CLINICAL TRIAL: NCT03394560
Title: Repetitive Transcranial Magnetic Stimulation Combined to Body Weight-support Treadmill Training in the Sensory-motor Recovery of Patients With Chronic Incomplete Spinal Cord Injury
Brief Title: rTMS and Body Weight-support Treadmill Training After Incomplete Spinal Cord Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Fernanda Natacha Rufino Nogueira, Bachelor in physical therapy, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rTMS_BWSTT_SCI
Record Dates: First submitted 2017-12-22; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; transcranial magnetic stimulation; body weight-support treadmill training; gait
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-frequency rTMS + BWSTT (Experimental): a randomized, sham-controlled, double-blinded and parallel group trial (12 therapeutic sessions) with the combination between body weight-support treadmill training combined and high-frequency rTMS in improving the sensory-motor function of adult patients with chronic incomplete thoracolumbar spinal cord injury. The sessions will be performed three times a week for a month.
  Interventions: Device: High frequency repetitive transcranial magnetic stimulation
- sham rTMS + BWSTT (Sham Comparator): a randomized, sham-controlled, double-blinded and parallel group trial (12 therapeutic sessions) with the combination between body weight-support treadmill training combined and high-frequency rTMS in improving the sensory-motor function of adult patients with chronic incomplete thoracolumbar spinal cord injury. The sessions will be performed three times a week for a month.
  Interventions: Device: Sham High frequency repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: High frequency repetitive transcranial magnetic stimulation — Gait training with body weight support will be performed through Biodex Rehabilitation treadmill. It will performed for 20 minutes and researchers will assist the patient in placing the foot on the ground, in the extension of the knee and in the alignment of pelvis and trunk. The percentage of body weight support and speed of treadmill will be modified based on the performance of each patient. Repetitive transcranial magnetic stimulation will be applied by an eight-shaped coil positioned on the patient's scalp and performed according to the 10-20 international system (primary motor cortex). In sham rTMS two coils will be used: (i) a coil connected to the stimulator will be positioned behind the patient (away from the scalp) to generate characteristic stimulus sound, and (ii) another coil will be disconnected from the stimulator and positioned on the scalp individual. The active and sham stimulation will last 20 minutes.
  Other Names: Body Weight-support Treadmill Training
  Arms: high-frequency rTMS + BWSTT
Device: Sham High frequency repetitive transcranial magnetic stimulation — Gait training with body weight support will be performed through Biodex Rehabilitation treadmill. It will performed for 20 minutes and researchers will assist the patient in placing the foot on the ground, in the extension of the knee and in the alignment of pelvis and trunk. The percentage of body weight support and speed of treadmill will be modified based on the performance of each patient. Repetitive transcranial magnetic stimulation will be applied by an eight-shaped coil positioned on the patient's scalp and performed according to the 10-20 international system (primary motor cortex). In sham rTMS two coils will be used: (i) a coil connected to the stimulator will be positioned behind the patient (away from the scalp) to generate characteristic stimulus sound, and (ii) another coil will be disconnected from the stimulator and positioned on the scalp individual. The active and sham stimulation will last 20 minutes.
  Other Names: Body Weight-support Treadmill Training
  Arms: sham rTMS + BWSTT

SUMMARY:
The aim of this study is to verify the efficacy of body weight-support treadmill training combined with high-frequency rTMS in improving the sensory-motor function of adult patients with chronic incomplete thoracolumbar spinal cord injury.

DETAILED DESCRIPTION:
A randomized, sham-controlled, double-blinded and parallel group trial (12 therapeutic sessions). Active or sham rTMS will be combined with body weight-support treadmill training to verify the improvement of sensory-motor function in patients with incomplete spinal cord injury. Behavioral assessments will be performed before, after 6 and 12 therapeutic sessions and at the 30-day follow-up after the intervention, though: (i) the WISCI-II Index; (ii) ASIA Impairment Scale (AIS), (iii) ASIA Lower Extremities Motor Scale (LEMS), (iv) Ashworth Modified Scale; (v) the Functional Independence Measure (SCIM-III), (vi) the Short Form Health Survey 36 (SF-36) and (vii) the Patient Global Impression of Change Scale - (PGICS).

ELIGIBILITY:
Inclusion Criteria:

* Presented clinical diagnostic of incomplete thoraco-lumbar spinal cord injury, provided by a neurologist (below the T1 level).
* Duration injury of at least 8 months.
* Presented degree of C or D according to the ASIA Impairment Scale (AIS) scale of the American Spinal Cord Injury Association.
* Patients who are not community walkers.

Exclusion Criteria:

* Pregnant women;
* Pacemaker;
* Historic of seizures;
* Metallic implants in the head;
* Patients with clinical evidence of brain injuries;
* Patients with neurological and / or orthopedic pathologies that have repercussion on a gait and the disadvantages
* Use of neuroleptic medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-30 (Estimated); Primary Completion 2018-08-30 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes on Walking Index for Spinal Cord Injury II (WISCI-II) | (i) Baseline - one day before the intervention, (ii) T0 - after 2 weeks, (iii) T1- after 4 weeks (iv) T2 - 1 month after the end of the intervention.
  this is international scale, designed to identify an improvement in the ability to perform gait with spinal cord injury under environmental conditions. The WISCI-II is considered standard for gait evaluation of patients with spinal cord injury inserted in clinical trials. The WISCI-II categorizes patients' ability to perform a gait on 20 different levels by considering the following: distance traveled, need for assistance, assistance from others people, and gait devices.
Changes on ASIA Impairment Scale (AIS) | (i) Baseline - one day before the intervention, (ii) T1- after 4 weeks and (iv) T2 - 1 month after the end of the intervention.
  this is international scale, it is the gold standard for the diagnosis of spinal cord injury and is used worldwide. The AIS categorizes the lesion from full spinal cord injury to normal degree, according to sensory-motor preservation, passing through 3 degrees of spinal cord injury (A , B, C, D or E).

SECONDARY OUTCOMES:
Changes on Spinal cord independence measure (Self-Reported) III (SCIM-III) | (i) Baseline - one day before the intervention, (ii) T1- after 4 weeks and (iv) T2 - 1 month after the end of the intervention
  The scale assesses patients' ability to perform tasks inherent to spinal cord injury and detects improvements in their functionality. The SCIM-III is a scale from 0 to 100 points and divides into three main domains: self-care (feeding, bathing, dressing and cleanliness), breathing, sphincter control and mobility (indoors and out home and transfers).
Change from Modified Ashworth scale (MAS) | (i) Baseline - one day before the intervention, (ii) T0 - after 2 weeks, (iii) T1- after 4 weeks (iv) T2 - 1 month after the end of the intervention.
  Modified Ashworth scale uses a 6-point scale to score the average resistance to passive for movement each joint. In this study, it will assess muscles: flexors and extensors hip, flexors and extensors knee, dorsiflexors and plantar flexors ankle.
Changes on Short-Form Health Survey (SF-36) | (i) Baseline - one day before the intervention, (ii) T1- after 4 weeks and (iv) T2 - 1 month after the end of the intervention
  The SF-36 is a multidimensional questionnaire consisting of 36 items, encompassed in eight scales or components: i. Functional capacity - 10 items, ii. Limitation by physical resources - 4 items, iii. Pain - 2 items, iv. General health status - 5 items, v. Vitality - 4 items, vi. Social Aspects - 2 items, vii. Limitation by emotional aspects - 3 items, viii. Mental Health - 5 items and one comparative question more for assessment between how current health conditions and a year ago.
Changes on Patient Global Impression of Change Scale - (PGICS) | (i)T0 - after 2 weeks, (ii) T1- after 4 weeks and (iii) T2 - 1 month after the end of the intervention.
  The PGICS is a one-dimensional measure in which individuals rate their improvement associated with intervention on a scale of 7 items ranging from "1 = no change" to "7 = Much better". This scale has already been validated in Brazil and has been used in clinical practice assays with spinal cord injury.
Changes on Lower Extremities Motor Scale (LEMS) from ASIA | (i) Baseline - one day before the intervention, (ii) T1- after 4 weeks and (iv) T2 - 1 month after the end of the intervention
  It is international scale, the LEMS is composed from the sum of muscle function grading of the five key muscles of the lower limbs (hip flexors, knee extensors, long toe extensors, ankle dorsiflexors and ankle plantar flexors) of ASIA. The score of each muscle can graded from "0" to "5" and the total LEMS score can graded from "0 to 50", for this, it should be added the score of the five muscles of each lower limb (left and right).

CONTACTS AND LOCATIONS:
Overall Officials: Lívia S Nascimento, MSc, Study Chair — Applied Neuroscience Laboratory; Marina Berenguer, PT, Study Chair — Applied Neuroscience Laboratory
Locations (1):
- Applied Neuroscience Laboratory, Recife, Pernambuco, Brazil